CLINICAL TRIAL: NCT02690571
Title: Pulmonary Effects of 100% Biodiesel Exhaust
Acronym: BD100Broncho
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Jenny Bosson, MD, PhD, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 184-31M
Record Dates: First submitted 2016-02-09; First posted 2016-02-24 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Inflammation
Keywords: Air Pollution; Biodiesel exhaust; Bronchoscopy; Metabolomics
MeSH Terms: conditions — Inflammation | interventions — Bronchoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filtered air exposure (Sham Comparator): One hour exposure to filtered air during intermittent exercise in controlled chamber, 6 hours after exposure bronchoscopy is performed.
  Interventions: Other: Bronchoscopy
- Biodiesel exhaust exposure (Experimental): One hour exposure to biodiesel exhaust (generated at same running conditions as earlier studies with diesel exhaust at approximate particle matter concentration 300 mcg/m3) during intermittent exercise in controlled chamber. Six hours after exposure bronchoscopy is performed.
  Interventions: Other: Bronchoscopy

INTERVENTIONS:
Other: Bronchoscopy — The bronchoscopy procedure was performed six hours after completion of the exposure session, with sampling of endobronchial mucosal biopsies, bronchial wash and bronchoalveolar lavage performed under topical anaesthesia.

SUMMARY:
Air pollution is a global environmental and health concern, contributing to onset and deterioration of respiratory and cardiovascular diseases. As climate change and dependence on diminishing fossil fuel supplies have taken center stage in political and scientific debates, renewable carbon-neutral fuels like biodiesel receive increasing attention. The most common biodiesel within the European Union, rapeseed oil methyl ester (RME) is perceived to be a "green fuel", as it is sustainable and of biological origin, and therefore is often predicted to be less harmful to human health. Whilst replacing petrodiesel with biodiesel may have advantageous ecological impacts, consequences to respiratory health remained largely unexplored.

The purpose of the current study is to evaluate whether inhalation of 100% RME biodiesel exhaust would result in an acute airway inflammatory response in healthy human subjects, as shown previously following exposure to petrodiesel exhaust.

ELIGIBILITY:
Inclusion Criteria:

Normal ECG

Normal Lung function

Normal Blood samples

Exclusion Criteria:

Smoking

Pre-existing metabolomic, respiratory and cardiovascular disease

Exposure to high levels of pollutants in occupation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cytokines in Bronchial wash (BW) | 6 hours
  Bronchial wash (BW) collected by bronchoscopy will be analyzed for cytokines (%).
Cell counts in Bronchial Wash | 6 hours
  Bronchial wash (BW) collected by bronchoscopy will be analyzed for inflammatory cell counts (cells/ml).

SECONDARY OUTCOMES:
Oxylipin Metabolomic profiling | Baseline, 2 hours, 6 hours, 24 hours
  Metabolomic testing done with mass spectrometry on blood samples, BW and BAL.
Inflammation in bronchoalveolar lavage (BAL) | 6 hour
  BAL collected by bronchoscopy will be analyzed for inflammatory markers, such as cell counts (cells/ml).
Inflammation in endomucosal biopsies | 6 hours
  Biopsies collected by bronchoscopy will be analyzed for inflammatory markers, such as cell counts (cells/mm2).

CONTACTS AND LOCATIONS:
Overall Officials: Jenny A Bosson, MD, PhD, Principal Investigator — Umeå University